CLINICAL TRIAL: NCT03458390
Title: Colon Irrigation Using HyGIeaCare as Prep for PillCam COLON Procedure
Brief Title: Use of a Colon Irrigation Device as a Preparation for a Colon Visualization Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HyGIeaCare, Inc. (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HGP-0005
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2019-06

CONDITIONS: Screening Colonoscopy

STUDY DESIGN:
Intervention Model Description: HyGIeaCare colon irrigation procedure and PillCam COLON procedure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HyGIeaCare and PillCam COLON (Experimental): Patient will receive the HyGIeaCare colon irrigation prior to their PillCam COLON procedure
  Interventions: Device: HyGIeaCare colon irrigation

INTERVENTIONS:
Device: HyGIeaCare colon irrigation — PillCam COLON for visualization of bowel lining
  Other Names: PillCam COLON

SUMMARY:
A prospective, single center, study to evaluate the effectiveness of the HyGIeaCare Prep when used in combination with the PillCam COLON; the hypothesis is that the HyGIeaCare Prep will be easier for the patients to tolerate, and the results will be as good as the existing oral preparation.

DETAILED DESCRIPTION:
Patients who agree to participate in the study will have their HyGIeaCare procedure and then will present to the PillCam COLON room, in the same suite for the PillCam COLON procedure.

The commercial preparations for the PillCam COLON procedure will be the same, except the HyGIeaCare procedure will replace the split polyethylene glycol-electrolyte solution preparation.

2-days prior:

* Normal diet
* 10 glasses of liquid

  1-day prior:
* Clear liquid diet all day
* Dulcolax 2 tabs at 2pm and 2 tabs at 8pm
* Nothing by mouth after midnight

Day of Procedure:

* 6am- Dulcolax 2 tabs
* 8am- HyGIeaCare Procedure
* 9am- ingest PillCam Colon
* 10am- ingest Reglan
* At small bowel detection, drink 10oz SUPREP and 32oz water
* 3hrs later- drink 10oz SUPREP and 32oz water
* 2hrs later- insert suppository
* 2hrs later- light meal

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for the PillCam COLON procedure

Exclusion Criteria:

-

HyGIeaCare:

1. Patient has any condition that, in the opinion of the investigator, may adversely affect the compliance or safety of the patient or would limit the patient's ability to complete the study
2. Patient is treated long-term with narcotics.
3. Patient does not have any of the contraindications listed below:

   1. Cardiac: Congestive heart failure (NYHA class III or IV or Ejection Fraction <50%)
   2. GastrointestinaI: Intestinal perforation, carcinoma of the rectum, Fissures or fistula, Severe hemorrhoids, Abdominal hernia, recent colon or rectal surgery, abdominal surgery
   3. Genitourinary: Renal insufficiency (CC < 60 ml/min/173m2), cirrhosis with ascites
   4. Abdominal surgery within the last 6 months
   5. Pregnancy

PillCam COLON:

1. Subject has dysphagia or any swallowing disorder
2. Subject has congestive heart failure
3. Subject has Diabetes type I.
4. Subject has had prior abdominal surgery other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
5. Subject has a cardiac pacemaker or other implanted electro medical device.
6. Subject has any allergy or other known contraindication to the medications used in the study
7. Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
8. Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, and incomplete colonoscopies due to obstructions or NSAID enteropathy.
9. Subject with gastrointestinal motility disorders
10. Subject has known delayed gastric emptying
11. Subject has any condition, which precludes compliance with study and/or device instructions.
12. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
13. Subject suffers from life threatening conditions
14. Subject currently participating in another clinical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-01-19 (Actual); Study Completion 2020-01-19 (Actual)

PRIMARY OUTCOMES:
Effectiveness of colon irrigation | Immediately after colon irrigation, PillCam COLON will be administered. A video will be taken of the procedure which will be used to measure the effectiveness of the colon irrigation.
  Effectiveness of the HyGIeaCare Prep will be measured using a 5-point scale to evaluate the visual quality of bowel cleanliness identified in the PillCam Colon video (Excellent, Good, Fair, Adequate, Poor).

SECONDARY OUTCOMES:
Evaluation of adverse events | To be evaluated the day of the procedure
  The CTCAE tool will be used to evaluate outcomes
Evaluation of patient satisfaction | To be evaluated on the day of the procedure
  A standardized questionnaire will be used to measure outcomes

CONTACTS AND LOCATIONS:
Overall Officials: David A Johnson, MD, Principal Investigator — Eastern Virginia Medical Center; William Stassen, MD, Principal Investigator — Austin Gastroenterology
Locations (1):
- HyGIeaCare Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Research outcomes will be evaluated by external statistician.

REFERENCES:
- [Background] Sommers T, Corban C, Sengupta N, Jones M, Cheng V, Bollom A, Nurko S, Kelley J, Lembo A. Emergency department burden of constipation in the United States from 2006 to 2011. Am J Gastroenterol. 2015 Apr;110(4):572-9. doi: 10.1038/ajg.2015.64. Epub 2015 Mar 24. PMID 25803399
- [Result] Singh G, Lingala V, Wang H, Vadhavkar S, Kahler KH, Mithal A, Triadafilopoulos G. Use of health care resources and cost of care for adults with constipation. Clin Gastroenterol Hepatol. 2007 Sep;5(9):1053-8. doi: 10.1016/j.cgh.2007.04.019. Epub 2007 Jul 10. PMID 17625982
- See also: Hydrotherapy compared with polyethylene glycol-electrolyte solution lavage and aqueous sodium phosphate as bowel preparation for elective colonoscopy: A prospective, randomized, single blinded trial — http://www.academia.edu/3514319/Title_HYDROTHERAPY_COMPAIRED_WITH_PEG-ES_LAVAGE_AND_AQUEOUS_SODIUM_PHOSPHATE_AS_BOWEL_PREPARATION_FOR_ELECTIVE_COLONOSCOPY_A_PROSPECTIVE_RANDOMIZED_SINGLE_BLINDED_TRIAL
- See also: Randomized trial comparing high volume rectal water irrigation with standard 4 liter split-dose polyethlene glycol-electrolyte solution preparation before colonoscopy — http://www.alliedacademies.org/articles/randomized-trial-comparing-high-volume-rectal-water-irrigation-with-standard-4-l-splitdose-peg-preparation-before-colonoscopy.pdf
- See also: HyGIeaCare® Preparation for Colonoscopy-A Technical Update for Success — http://www.hygieacare.com/assets/2016_gagneja_hygieacare-preparation-for-colonscopy---a-technical-update-for-success.pdf
- See also: Multi-Dimensional Gastrointestinal Symptom Severity Index: Validation of a Brief GI Symptom Assessment Tool — https://link.springer.com/article/10.1007%2Fs10620-015-3647-3